CLINICAL TRIAL: NCT06739083
Title: Preparation and Evaluation of a Web-Based E-Mentoring Program for Newly Hired Nurses
Brief Title: E-Mentoring Program for Newly Hired Nurses
Acronym: E-Mentoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merve BEKE (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Merve BEKE, MSc, Registered Nurse, PhD Candidate, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 323S169; TUBİTAK (Other: The Scientific and Technological Research Council of Türkiye)
Record Dates: First submitted 2024-11-12; First posted 2024-12-18 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Healthy; Nurse
Keywords: e-mentoring; nurse; newly hired nurse; mentor; mentee

STUDY DESIGN:
Intervention Model Description: This study is designed as a single-group study consisting of both mentors and mentees.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- e-mentoring program (Experimental): The e-mentoring program is planned to last four weeks to facilitate the adaptation process of newly recruited nurses in intensive care units via the e-mentoring website.
  Interventions: Other: e-mentoring program

INTERVENTIONS:
Other: e-mentoring program — The e-mentoring program is planned to last four weeks to facilitate the adaptation process of newly recruited nurses in intensive care units via the e-mentoring website.

SUMMARY:
The E-mentorship Program is planned to last four weeks to facilitate the adaptation process of newly hired nurses in intensive care units. The program will be conducted through a specialized web-based e-mentorship platform, enabling experienced nurses to mentor and support the professional development of new hires.

This study aims to design, implement, evaluate and determine the effect of an e-mentorship program that will provide online support to facilitate the adaptation of new nurses to work.

Research Hypotheses H1 - The work readiness score of mentees who participated in the e-mentorship program is higher after the program than before the program.

H2 - The satisfaction with the use of the e-mentorship website is proportional to the work readiness score of mentees.

H3 - The design and usability of the e-mentorship website are effective in facilitating the adaptation of new nurses to work.

Research Goals

* Design of an e-mentoring program that nurses can use,
* Implementation of the e-mentoring program,
* Evaluation of the satisfaction of using the e-mentoring website,
* Determining the effect of job adaptation of new nurses.

DETAILED DESCRIPTION:
In Turkey, the adaptation of newly hired nurses to institutions and organizational culture typically occurs through an apprentice-mentor relationship under the guidance of experienced nurses. Within mentoring and guidance programs established by institutions, newly hired nurses work with mentors assigned by the organization. Mentors are expected to be continuously available to support new nurses, facilitate their learning processes, and foster adaptation to the work environment through constructive and critical guidance. However, in these programs, mentors often struggle to fulfill these responsibilities in addition to their daily tasks, finding it challenging to allocate time for their mentees and facing increased workloads; mentees, in turn, may have difficulty reaching their mentors when needed. Studies indicate that nurses participating in mentorship programs demonstrate lower turnover rates compared to those without such programs, underscoring the importance of mentorship.

Research on mentoring nurses in their first year of practice shows that mentorship reduces turnover, eases adaptation, and helps them develop essential professional skills. Mentors serve as role models for mentees and play a crucial role in fostering a supportive workplace culture. Furthermore, mentorship has been shown to reduce clinical practice-related stress. The findings from these studies highlight the effectiveness of mentorship programs in supporting the adaptation of new employees, while also emphasizing the need to eliminate time and space limitations for an effective mentoring process. These findings point to the potential benefits of e-mentorship. Leveraging emerging technologies is thus essential in facilitating the adaptation of newly hired nurses and fostering a skilled workforce. Notably, the literature does not currently include an e-mentorship application specifically for newly hired nurses in Turkey. This study aims to develop, implement, and evaluate an e-mentorship program, presenting an innovative contribution to the literature and holding significant potential for enhancing professional practice.

ELIGIBILITY:
Inclusion Criteria:

* Newly hired nurses (mentees) employed for less than one year
* Senior nurses (mentors) with at least three years of experience working in an adult intensive care unit
* Working as a nurse in a secondary or tertiary adult intensive care unit
* A minimum of a bachelor's degree in nursing for mentors (preferably a graduate degree)
* Possession of an intensive care nursing certification for mentors
* Possession of a smartphone with an operating system such as iOS or Android, or regular access to a computer

Exclusion Criteria:

* Failure to complete the e-mentoring program
* Currently employed for more than one year (for newly hired nurses/mentees)
* Less than three years of experience in an adult intensive care unit (for senior nurses/mentors)
* Lack of required nursing certifications or educational qualifications (for mentors)
* Inability to regularly access a smartphone with iOS/Android or a computer
* Currently on extended leave (e.g., maternity, medical, or personal leave)
* Participation in any other formal mentoring or similar professional development programs during the study period

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
The Work Readiness | At the beginning of the study and at study completion (an average of 6 months)
  The Work Readiness Scale, developed to assess the job readiness of newly hired nurses, consists of 46 items and four subscales (job competence, social intelligence, organizational awareness, personal work characteristics) and uses a 10-point Likert scale. Items are scored from 1 (strongly disagree) to 10 (strongly agree), with a minimum score of 46 and a maximum of 460, where higher scores indicate higher job readiness among newly hired nurses.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The intention to share individual participant data (IPD) will be carefully considered and determined in alignment with ethical guidelines and privacy regulations. Given the sensitive nature of the data collected in this study, particularly related to healthcare professionals' personal and professional characteristics, any decision to share IPD will involve ensuring participant confidentiality and complying with relevant data protection laws, including informed consent agreements. Should the IPD be shared, it will be made available only to researchers with appropriate ethical approvals and for purposes directly related to advancing scientific knowledge in the field. The data sharing plan will be clearly outlined and shared with participants in the informed consent process, with a commitment to safeguarding their rights and privacy. The final decision will be made upon review of the data's sensitivity and the potential benefits of sharing it with the wider research community.

REFERENCES:
- [Background] Baldwin A, Mills J, Birks M, Budden L. Reconciling professional identity: A grounded theory of nurse academics' role modelling for undergraduate students. Nurse Educ Today. 2017 Dec;59:1-5. doi: 10.1016/j.nedt.2017.08.010. Epub 2017 Sep 5. PMID 28898727
- [Result] Mansour M, Mattukoyya R. A Cross-Sectional Survey of British Newly Graduated Nurses' Experience of Organization Empowerment and of Challenging Unsafe Practices. J Contin Educ Nurs. 2018 Oct 1;49(10):474-481. doi: 10.3928/00220124-20180918-08. PMID 30257031
- [Result] Latham CL, Hogan M, Ringl K. Nurses supporting nurses: creating a mentoring program for staff nurses to improve the workforce environment. Nurs Adm Q. 2008 Jan-Mar;32(1):27-39. doi: 10.1097/01.NAQ.0000305945.23569.2b. PMID 18160861
- [Result] Chen CM, Lou MF. The effectiveness and application of mentorship programmes for recently registered nurses: a systematic review. J Nurs Manag. 2014 May;22(4):433-42. doi: 10.1111/jonm.12102. Epub 2013 Jul 15. PMID 23848442
- [Result] Zhang Y, Qian Y, Wu J, Wen F, Zhang Y. The effectiveness and implementation of mentoring program for newly graduated nurses: A systematic review. Nurse Educ Today. 2016 Feb;37:136-44. doi: 10.1016/j.nedt.2015.11.027. Epub 2015 Dec 12. PMID 26725949